CLINICAL TRIAL: NCT01328795
Title: Cardiogoniometry Zur Früherkennung Akuter Myokardischämien Bei ACS-Symptomatik
Brief Title: Cardiogoniometry (CGM) for Early Diagnosis of Acute Coronary Syndromes (ACS)
Acronym: CGM@ACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stiftung Institut fuer Herzinfarktforschung (Other)
Responsible Party: Prof. Jochen Senges, Institut für Herzinfarktforschung Ludwigshafen an der Universität Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CGM@ACS
Record Dates: First submitted 2011-02-11; First posted 2011-04-05 (Estimated); Last update posted 2011-04-05 (Estimated); Status verified 2011-04

CONDITIONS: Chest Pain
Keywords: Cardiogoniometry; Chest Pain Unit; ST-elevation; Troponin; Catheter intervention; Fast Track
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: cardiogoniometry — In the course of the project a cardiogoniometry will be carried out during the ambulant or residential hospitalization before the coronary angiography.

SUMMARY:
Aims of the study:

Patients in a Chest Pain Unit (CPU) are examined to clarify if the cause of pain is cardiac or not. To identify patients with ST-elevation and other electrocardiogram (ECG) modifications a normal 12-lead ECG is used. The diagnosis non-st-elevation myocardial infarction is determined with the help of the ischemic marker Troponin. However, Troponin levels are elevated earliest 3 to 4 hours after the ischemic event, so that a negative Troponin result at the time of hospital admission is insufficient. Thus the guidelines of the German Society of Cardiology demand a second measurement after 6 to 12 hours. In rare cases false positive Troponin levels have been reported (e.g. in patients with renal insufficiency).

The aim of this study is to determine if in the early phase of diagnostic assessment cardiogoniometry can improve differentiation between patients with cardiac (ischemic) emergency and patients with non-cardiac (non-ischemic) cause of pain. Furthermore it will be evaluated if cardiogoniometry is capable to diagnose patients with non-ST-elevation myocardial infarction (NSTEMI) to the same extent as Troponin. This could avoid time loss until a possibly necessary catheter intervention ("fast track").

To clarify these questions the result of the cardiogoniometry will be compared with the leading diagnosis of the Chest Pain Unit, the diagnosis at hospital discharge as well as with the angiographic findings (as a gold standard). Therefore the performance of cardiac catheterization within 72 hours after start of symptoms is a mandatory inclusion criterion.

DETAILED DESCRIPTION:
The cardiogoniometry vectorcardiography is a procedure that allows a stress-free and non-invasive diagnosis of myocardial ischemia: five thoracic electrodes as well as the heart flow in orthogonal summation vectors are recorded by a computer-assisted method in three dimensions.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* thoracic pain, or pain radiating to neck or arm, or acute dyspnoea
* coronary angiography within 72 hours after start of symptoms

Exclusion Criteria:

* ST elevation myocardial infarction
* hemodynamically unstable patients, provided that the application of CGM may lead to an unacceptable delay in diagnosis and therapy
* lack of blood samples for troponin determination at admission
* patients with cardiac pacemaker
* cardiogenic shock
* tachycardia (HR > 100)
* > 50% extra systoles
* branch block
* atrial fibrillation
* no informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2009-06; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Difference between cardiogoniometry finding and leading diagnoses of chest pain unit, coronary angiography, and at discharge in assessing the origin of chest pain | 72 hours
  Aim is to examine if cardiogoniometry can provide additional information for the decision to perform a diagnostic coronary angiography and if so, which additional value it has. To assess the value of cardiogoniometry its results are compared with the leading diagnosis of the Chest Pain Unit, the diagnosis at hospital discharge as well as with the angiographic findings (as a gold standard).

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Senges, MD, Study Director — Stiftung Institut fuer Herzinfarktfoschung